CLINICAL TRIAL: NCT05667779
Title: A Randomized, Placebo-Controlled, Double-blind, Single Ascending Dose, First in Human Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of QRL-101 in Healthy Participants
Brief Title: A Study Evaluating Safety, Tolerability, and Pharmacokinetics of QRL-101 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QurAlis Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QRL-101-01; 2022-002484-30 (EudraCT Number)
Record Dates: First submitted 2022-12-19; First posted 2022-12-29 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, double-blind, placebo-controlled single ascending dose (SAD) study in healthy participants with the primary goal of evaluating the safety and tolerability of QRL-101.
Who Masked: Participant, Investigator
Masking Description: A participant and investigator-blinded, randomized, placebo-controlled design will be used to minimize bias in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- QRL-101 (Experimental): Single-ascending doses of QRL-101 will be administered orally to healthy participants
  Interventions: Drug: QRL-101
- Placebo (Placebo Comparator): Single-ascending doses of comparator placebo will be administered orally to healthy participants
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: QRL-101 — Single-ascending doses of QRL-101 will be orally administered. The dose levels may change subject to available nonclinical, clinical, safety, and PK data.
  Arms: QRL-101
Other: Placebo — A placebo comparator will be administered at all dose levels.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of ascending single doses of QRL-101 in male and female healthy participants. The findings from this study will be used to inform the development of QRL-101 for people living with ALS.

DETAILED DESCRIPTION:
Phase 1, single-site study to evaluate the safety, tolerability, and pharmacokinetics (PK) of ascending single doses of QRL-101 administered orally in healthy male and female participants. Up to 16 cohorts of 8 participants each, randomized 6:2 (QRL-101: placebo) will be tested. The approximate total duration of study participation for each participant may be up to 40 days.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age 18 to 70 years of age inclusive at the time of signing the informed consent.
2. Clinical chemistry laboratory values within acceptable range for the population, as per investigator judgment.
3. Body mass index of 18 to 32 kg/m2 (inclusive).
4. Willing and able to practice effective contraception.

EXCLUSION CRITERIA

1. Currently enrolled in any other clinical trial involving a study drug or off-label use of a drug or device, or any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Any participant in >4 studies a year and/or has participated in a clinical trial within 1 month of expected dosing date.
3. History or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric, or neurological disease, convulsions, or any clinically significant laboratory abnormality that, in the judgment of the investigator, indicate a medical problem that would preclude study participation.

*Other inclusion and exclusion criteria may apply*

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more treatment emergent adverse events and serious adverse events. | Baseline through Follow up (Day 10)
  Endpoints: A summary of treatment emergent adverse events (AEs), serious adverse events (SAEs), and other non-serious adverse events, regardless of causality, will be reported in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Pharmacokinetics (plasma): Maximum observed concentration of QRL-101 | Baseline through Follow up (Day 10)
  Endpoint: Maximum observed concentration (Cmax) of QRL-101
Pharmacokinetics (plasma): Area under the concentration time curve from 0 to 24 h (AUC 0-24h) of QRL-101 | Baseline through Follow up (Day 10)
  Endpoint: Area under the concentration time curve from zero to infinity (AUC 0-24h) of QRL-101
Pharmacokinetics (plasma): Time of maximum concentration of QRL-101 | Baseline through Follow up (Day 10)
  Endpoint: Time of maximum concentration (Tmax) of QRL-101

CONTACTS AND LOCATIONS:
Overall Officials: Salah Hadi, MD, Principal Investigator — ICON plc
Locations (1):
- ICON plc. Van Swietenlaan 6, Groningen, Netherlands